CLINICAL TRIAL: NCT02117310
Title: Proposal for Intraoperative Administration of Intravenous Indocyanine Green to Evaluate Sphenopalatine Artery Location and Patency in Harvesting and Positioning a Pedicled Nasoseptal Mucosal Flap in Endoscopic Endonasal Cranial Base Surgery
Brief Title: ICG Use in Angiography for Nasoseptal Flap Harvest
Acronym: ICG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel Prevedello, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013H0414
Record Dates: First submitted 2014-03-20; First posted 2014-04-17 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Skull Base Neoplasms
MeSH Terms: conditions — Skull Base Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG (Experimental): Angiography with administered ICG
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — ICG will be administered to identify the blood supply at two distinct stages of endonasal cranial base surgery: during nasoseptal flap harvest and after final positioning of the nasoseptal flap to ensure its viability before ending the case.

SUMMARY:
This is a feasibility study in which indocyanine green (ICG) will be administered during routine expanded endonasal approach (EEA) for cranial base pathologies in which a nasoseptal flap harvest will be necessary. The research entails administering ICG, which is already widely used during open neurosurgical procedures, to identify the blood supply at two distinct stages of endonasal cranial base surgery: during nasoseptal flap harvest and after final positioning of the nasoseptal flap to ensure its viability before ending the case.

DETAILED DESCRIPTION:
This study is being done to determine if it is feasible to use angiography during endo-nasal surgery. During the angiography indocyanine green (ICG) will be injected into the patients IV tubing to help see the arteries. ICG is routinely used in vascular surgeries on the brain but not for endo-nasal surgery. The purpose of this study is to see how well intraoperative angiography using ICG can be done during endonasal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Patients undergoing an EEA for cranial base pathology that may require nasoseptal flap harvest

Exclusion Criteria:

* History of sulfa, iodide, or penicillin allergy
* Pregnant or breast feeding
* Preoperative lack of indication for nasoseptal flap harvest
* Previous anaphylactic reaction to ICG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Prevedello, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ICG-Angiography With Administered ICG: Indocyanine green: ICG will be administered to identify the blood supply at two distinct stages of endonasal cranial base surgery: during nasoseptal flap harvest and after final positioning of the nasoseptal flap to ensure its viability before ending the case.
Period: Overall Study
Arm/Group | ICG-Angiography With Administered ICG
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ICG-Angiography With Administered ICG
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 41.4 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which Angiograghy is Used to Visualize Nasoseptal Mucosa Better Than What is Done Standard of Care in This Surgery.
Description: The researcher will administer ICG, which is already widely used during open neurosurgical procedures, to identify the blood supply at two distinct stages of endonasal cranial base surgery: during nasoseptal flap harvest and after final positioning of the nasoseptal flap to ensure its viability before ending the case. This study will determine feasibility of other larger clinical trials using this method.
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | ICG-Angiography With Administered ICG
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Arm/Group | ICG-Angiography With Administered ICG
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No